CLINICAL TRIAL: NCT05957159
Title: Investigating the Mu:Kappa Opioid Receptor Imbalance in Alcohol Use Disorder
Acronym: Mu Kappa
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kelly Cosgrove, Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000035344; 1R01AA030528-01A1 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-07-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Alcohol cessation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: All subjects will be asked to complete both PKAB and CFN PET Imaging scans, AUD subset will participate in a detoxification program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Use Disorder population completing Detoxification (Experimental): Subjects will be asked to complete both 90 minute [11C]CFN and 90 minute [11C]PKAB PET Imaging after 1-3 days of a detoxification program.
  Interventions: Other: Detoxification Program; Radiation: PKAB; Radiation: CFN
- Healthy Control population (Experimental): Subjects will be asked to complete both a 90 minute [11C]CFN and a 90 minute [11C]PKAB PET Imaging.
  Interventions: Radiation: PKAB; Radiation: CFN

INTERVENTIONS:
Other: Detoxification Program — Patients will begin inpatient or outpatient detoxification prior to completing imaging
  Arms: Alcohol Use Disorder population completing Detoxification
Radiation: PKAB — 90 PET Imaging Scan using [11C]LY2795050 (AKA [11C]PKAB)
Radiation: CFN — 90 Pet Imaging Scan using [11C]-Carfentanil

SUMMARY:
The primary objective of this multimodal positron emission tomography (PET) study is to use PET brain imaging to measure both MOR (Mu-Opioid receptors) and KOR (kappa-opioid receptors) in participants with alcohol use disorder (AUD) and to quantify the relationships between MOR and KOR, separately and jointly, to key clinical outcomes (e.g., craving, mood, withdrawal, time to lapse) during a quit attempt.

DETAILED DESCRIPTION:
Primary Objective

The primary objective of this multimodal positron emission tomography (PET) study is to use PET brain imaging to measure both MOR (Mu-Opioid receptors) and KOR (kappa-opioid receptors) in participants with alcohol use disorder (AUD) and to quantify the relationships between MOR and KOR, separately and jointly, to key clinical outcomes (e.g., craving, mood, withdrawal, time to lapse) during a quit attempt. Investigators will achieve this goal by completing the following aims:

Aim 1: To determine whether participants with AUD in early abstinence (up to 6 days) have altered MOR and KOR availability compared to healthy subjects. Investigators propose to recruit 50 people with AUD (DSM-5 diagnosis) and 50 age- and sex-matched controls to each participate in one [11C]CFN and one [11C]PKAB PET scan. Participants with AUD will participate either 1) in a medically supervised inpatient unit, the Clinical Neuroscience Research Unit (CNRU), for ~6 days, or 2) will stop drinking on an outpatient basis with daily meetings for ~6 days. Measures of craving (including a cue reactivity task), mood, withdrawal, and drinking outcomes will be collected. Hypothesis: participants with AUD will have significantly higher MOR in ventral striatum, but lower KOR in amygdala and whole striatum compared to control participants.

Aim 2: To relate measures of MOR and KOR availability to clinical outcomes during early and late abstinence. Early abstinence (~6 days) will be followed by an outpatient quit attempt for an additional 3 weeks supported by contingency management. Measures of craving, mood, withdrawal, and drinking outcomes will be collected throughout the study. Hypothesis: Taken one at a time, MOR availability in ventral striatum as well as KOR in the amygdala and whole striatum will each be significantly associated with abstinence-induced craving, mood, withdrawal, and time to lapse in participants with AUD.

Aim 3: To maximize use of neuroimaging data via machine-learning-based clustering to identify biomarkers of the joint (MOR, KOR) dataset that characterize clinical outcomes in AUD during a quit attempt. Primary. The investigators will determine whether clusters of AUD patients based on features of the joint (MOR, KOR) data are significantly associated with distinct clinical outcomes (e.g., time to lapse) during a quit attempt. Secondary. Investigators will test the classification accuracy of our clustering approach. Hypotheses: Clustering of joint (MOR, KOR) data will yield clusters of AUD patients with significantly different clinical responses to a quit attempt. Clusters will be more compact (distinct) than if based on demographics or a single type of PET image, alone. A classification scheme based on (MOR, KOR) data will assign individual patients to pre-defined clusters with high classification accuracy, that is, to the cluster that best reflects their clinical outcomes.

Aim 4: To determine whether MOR and KOR availability normalizes over the course of abstinence. Subjects who do not drop out of the study in the first 3 weeks may return for one [11C]CFN, one [11C]PKAB PET scan, and one MRI during weeks 3-6 of the study. This will allow us to gain information on the changes in the MOR and KOR systems that occur during a quit attempt. Investigators hypothesize a reduction in MOR and increase in KOR within subject in participants who are able to maintain abstinence.

Secondary Objective (if applicable) The secondary objective of this study is to evaluate the predictive ability of the clustering method, i.e., its potential for personalized prediction of individual clinical outcomes. For any 'new' subject not used for the initial clustering, investigators will assign it to a cluster by a K-nearest neighbor approach.

ELIGIBILITY:
Inclusion Criteria:

* Participants with AUD will have a current diagnosis of AUD according to DSM-5 criteria (i.e., SCID-5 ascertained diagnosis, confirmed by the Principal Investigators);
* Participants with AUD will meet the following drinking criteria: males will drink > 14 drinks per week and exceed 4 drinks per day at least twice per week; females will drink > 7 drinks per week and exceed 3 drinks per day at least twice per week. They must meet drinking criteria during a consecutive 30-day period within the 90 days prior to intake;
* Participants with AUD will indicate willingness to abstain from alcohol and engage in a quit attempt;
* Healthy subjects will have no current or past diagnosis of AUD or other significant substance use disorder. They will drink less than 5 alcoholic drinks per week with no heavy drinking days (i.e., >4 drinks/day for men; >3 drinks/day for women) in the last 30 days;
* Able to read and write English and to provide voluntary, written informed consent;
* Agree to have blood drawn for genotyping of the OPRM1 which has been shown to impact the [11C]CFN outcome measure, BPND50.

Exclusion Criteria:

* Current significant medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology that would impact the integrity of the data (note that elevated liver enzymes for individuals with AUD will not be exclusionary);
* Past or current neurological disorder or disorders affecting the brain including but not limited to multiple sclerosis, history of stroke, brain tumors, traumatic brain injury with loss of consciousness, seizure disorder;
* Current significant psychiatric disorder including severe substance use disorder (other than alcohol or tobacco use disorders*), and past or current psychotic symptoms;
* Regular use in the past 6 months of any prescription, psychoactive or herbal medications (e.g., antidepressants, antipsychotics, anxiolytics) that would impact the integrity of the data (e.g., naltrexone); No subject will be asked to stop taking medication to participate in the study;
* Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or her partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD;
* Contraindications to MRI such as claustrophobia or metal in their body;
* Subjects whose participation would cause them to exceed yearly radiation limits for research subjects

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Regional binding availability and volume of distribution of (Mu-Opioid receptors) | Within first 6 days of abstinence
  Time activity curves will be extracted from brain regions of interest during [11C]CFN PET Imaging. AUD subjects will be asked to complete this within first 6 days of abstinence. Healthy control subjects will be matched based on sex(Male/Female), smoking status (current/former/nonsmoker), and BMI (kg/m^2)
Regional binding availability and volume of distribution of (Mu-Opioid receptors) | Between 3 to 6 weeks into alcohol cessation
  Time activity curves will be extracted from brain regions of interest during [11C]CFN PET Imaging. AUD subjects will be asked to complete this 3 -6 weeks into alcohol cessation. Healthy control subjects will be matched based on sex(Male/Female), smoking status (current/former/nonsmoker), and BMI (kg/m^2)
Regional binding availability and volume of distribution of (Kappa-Opioid receptors) | Within first 6 days of abstinence
  Time activity curves will be extracted from brain regions of interest during [11C]PKAB PET Imaging. AUD subjects will be asked to complete this within first 6 days of abstinence. Healthy control subjects will be matched based on sex(Male/Female), smoking status (current/former/nonsmoker), and BMI (kg/m^2)
Regional binding availability and volume of distribution of (Kappa-Opioid receptors) | Between 3 to 6 weeks into alcohol cessation
  Time activity curves will be extracted from brain regions of interest during [11C]PKAB PET Imaging. AUD subjects will be asked to complete this 3 -6 weeks into alcohol cessation. Healthy control subjects will be matched based on sex(Male/Female), smoking status (current/former/nonsmoker), and BMI (kg/m^2)
Alcohol Cue Reactivity Craving | Within first 6 days of abstinence
  Investigators will follow the paradigm developed for the NIAAA Human Laboratory Medication Screening Program (HLAB). In the paradigm, participants will be first exposed to a glass of water and then to their typical alcoholic beverage, separated by a 90 second rest period. They will be instructed to not drink but to sniff the beverages for a fixed duration. Immediately after, alcohol craving and beverage liking will be assessed. AUD subjects will be asked to complete this within first 6 days of abstinence. Healthy control subjects will be matched based on sex(Male/Female), smoking status (current/former/nonsmoker), and BMI (kg/m^2)
Change in Alcohol Withdrawal | Up to 1 month prior to initial imaging and up to 6 days into alcohol cessation
  Withdrawal will be assessed using The Clinical Institute Withdrawal Assessment (CIWA-R)64. AUD and Healthy controls will be asked to complete this paper questionnaire up to 1 month prior to CFN and PKAB PET Imaging and once again up to 6 days into alcohol cessation for AUD population
  Range: 0- 67, higher scores indicating more symptoms of withdrawal.
Change in Alcohol Use | Up to 1 month prior to initial imaging and up to 6 days into alcohol cessation
  Assessed using the TimeLine Followback (TLFB)62 and BACtrack Skyn; AUD and Healthy controls will be asked to complete this paper questionnaire up to 1 month prior to CFN and PKAB PET Imaging and once again up to 6 days into alcohol cessation for AUD population.
  Calendar style open ended.
  Minimum 0 alcohol uses in past month -31 sittings of alcohol in past month
Change in Alcohol Craving | Up to 1 month prior to initial imaging and up to 6 days into alcohol cessation
  Craving will be assessed with Alcohol Craving Scale (ACS, adapted from Singleton et al.63),
  Range: 47 to 329, higher scores indicate higher craving to alcohol
Change in Mood | Up to 1 month prior to initial imaging and up to 6 days into alcohol cessation
  Mood, anhedonia symptoms will be assessed with the Center for Epidemiologic Studies Depression Scale (CES-D) Range : 0 to 60. Higher scores indicate more symptoms of depression.

SECONDARY OUTCOMES:
Baseline Verbal Memory | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  Cogstate International Shopping List Task - a computerized task to assess verbal learning and memory.
  # of correctly recalled items from a grocery list (3 trials). Verbal Recalled item from grocery list after delay (1 trial; higher ~better memory/recall)
  Range: up to 0 to 36 errors (per trial), up to 108 errors for all 3 trials.
Baseline Verbal Memory | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  Cogstate International Shopping List Task - a computerized task to assess verbal learning and memory.
  # of correctly recalled items from a grocery list (3 trials). Verbal Recalled item from grocery list after delay (1 trial; higher ~better memory/recall)
  Range: 0 to 36 errors (per trial), up to 108 errors for all 3 trials.
Baseline Executive Function | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  : Cogstate Groton Maze Learning Task - a computerized task to assess executive function and spatial problem solving. # of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function.
  Range: 0-140 errors per trial, 0- 700 errors for all five trials
Test Executive Function | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  : Cogstate Groton Maze Learning Task - a computerized task to assess executive function and spatial problem solving. # of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function.
  Range: 0-140 errors per trial, 0- 700 errors for all five trials
Baseline Visual Processing Speed | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  Cogstate Detection Task - a computerized task to assess psychomotor function and speed of processing. Visual -motor processing speed: response latency to detect a card flipped over (log10(ms); higher~ worse processing speed).
  Range: 0 milliseconds - 30 minute times out.
Test Visual Processing Speed | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  Cogstate Detection Task - a computerized task to assess psychomotor function and speed of processing. Visual -motor processing speed: response latency to detect a card flipped over (log10(ms); higher~ worse processing speed).
  Range: 0 milliseconds - 30 minute times out.
Baseline Visual Attention | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  Identification Task - a computerized task to assess visual attention and vigilance. Response latency to identify card color (log10(ms)higher ~worse attention)
  Range: 0 milliseconds - 30 minute times out.
Test Visual Attention | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  Identification Task - a computerized task to assess visual attention and vigilance. Response latency to identify card color (log10(ms)higher ~worse attention)
  Range: 0 milliseconds - 30 minute times out.
Baseline Visual Learning | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  One Card Learning Task - a computerized task to assess visual learning and memory. Visual Learning: % of correctly identified repeat cards (arcsine% correct); higher ~ better learning.
  Range: 66-88 cards
Test Visual Learning | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  One Card Learning Task - a computerized task to assess visual learning and memory. Visual Learning: % of correctly identified repeat cards (arcsine% correct); higher ~ better learning.
  Range: 66-88
Baseline Working Memory One Back | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  One Back Task - computerized tasks to assess attention and working memory. Working memory: % of correctly identified cards that matched the card presented either one card previously (arcsine(% correct); Higher~ better working memory
  Range: ONB 24-31,
Test Working Memory One Back | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  One Back Task - computerized tasks to assess attention and working memory. Working memory: % of correctly identified cards that matched the card presented either one card previously (arcsine(% correct); Higher~ better working memory
  Range: ONB 24-31
Baseline Working Memory Two Back | Up to 3 months prior to initial imaging or on initial imaging day (depending hospital availability
  One Back Task - computerized tasks to assess attention and working memory. Working memory: % of correctly identified cards that matched the card presented either one card previously (arcsine(% correct); Higher~ better working memory
  Range: Two Back 24-32
Test Working Memory Two Back | Completed on second PKAB/CFN imaging day (Between 3 to 6 weeks into alcohol cessation)
  Two Back Task - computerized tasks to assess attention and working memory. Working memory: % of correctly identified cards that matched the card presented either one card previously (arcsine(% correct); Higher~ better working memory
  Range: Two Back 24-32

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No